CLINICAL TRIAL: NCT05227937
Title: Single Dose Amikacin for Uncomplicated Cystitis in the Emergency Department (ED): A Feasibility Study
Brief Title: Single Dose Amikacin for Uncomplicated Cystitis in the ED: A Feasibility Study
Status: Recruiting | Type: Observational
Sponsor: Antonios Likourezos (Other)
Responsible Party: Sponsor-Investigator, Antonios Likourezos, Research Administration Director, Maimonides Medical Center
Organization: Maimonides Medical Center (Other)
Other Study IDs: 2021-07-07
Record Dates: First submitted 2022-01-27; First posted 2022-02-08 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Urinary Tract Infections
Keywords: urinary tract infections; amikacin; emergency medicine
MeSH Terms: conditions — Urinary Tract Infections | interventions — Amikacin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Single Dose Amikacin: Patient will be treated with amikacin 15 mg/kg IV or IM, based on actual body weight; for patients >120% of IBW, we will use AdjBW (IBW + 0.4(ABW-IBW)) rounded to nearest 50 mg. Patients who already have an IV will receive the medication IV, otherwise the dose will be given IM.
  Interventions: Drug: Amikacin

INTERVENTIONS:
Drug: Amikacin — patient will be treated with amikacin 15 mg/kg IV or IM, based on actual body weight; for patients >120% of IBW, we will use AdjBW (IBW + 0.4(ABW-IBW)) rounded to nearest 50 mg. Patients who already have an IV will receive the medication IV, otherwise the dose will be given IM.

SUMMARY:
The purpose of this study is to determine if a single dose of amikacin (a type of antibiotic) can be used to effectively treat emergency department patients with uncomplicated cystitis (inflammation of the bladder). Participating in this study will allow the patient to treat their urinary tract infection (UTI) with a single intramuscular (IM (into the arm)) or intravenous (IV (into the vein)) shot of amikacin, rather than having to go to the pharmacy to pick up a prescription for antibiotics, and then take antibiotics for 3-7 days. A single dose of amikacin has been demonstrated to be safe, effective and well tolerated in other studies, but some patients may decline to participate because they do not wish to have an IV or IM shot, or because they don't want to speak on the phone with a research assistant three times over the next 30 days.

DETAILED DESCRIPTION:
he study is a prospective open-label cohort study that seeks to enroll 75 ED patients diagnosed with uncomplicated cystitis. Enrolled patients will be treated with a single dose of amikacin. The primary endpoint is clinical cure at 3 days. We chose a non-comparative design as our treatment strategy is literature- and guideline- supported; our goal is demonstrate that it is feasible to execute this approach out of the emergency department. Urine culture is not recommended in the in the initial management of patients with uncomplicated UTI treated in emergency or primary care settings.3

Data Collection Procedures: Patients will be enrolled as a convenience sample by the research team. The investigators will determine eligibility, approach the ED clinical team, then approach and consent the patient.

If consented, patient will be treated with amikacin 15 mg/kg IV or IM, based on actual body weight; for patients >120% of IBW, we will use AdjBW (IBW + 0.4(ABW-IBW)) rounded to nearest 50 mg. Patients who already have an IV will receive the medication IV, otherwise the dose will be given IM.

The study measurements at enrollment are age, PMH, meds, allergies, symptoms, and symptom duration as well as urinalysis results, amikacin dose and route. Telephone follow-up at 3, 7, and 30 days will include the following data points: symptom resolution: (complete resolution / mostly better / a little better / same / worse); any new symptoms; any provider visits since index visit (if any visits, describe).

ELIGIBILITY:
Inclusion Criteria:

* female emergency medicine patients
* ≥14 years of age
* uncomplicated urinary tract infection
* a primary urinary complaint and nitrite-positive urine.

Exclusion Criteria:

* pregnancy
* abnormal genitourinary tract
* recent urinary tract instrumentation
* immunosuppression
* CrCl < 25 mL/min
* evidence of pyelonephritis or sepsis
* any antibiotic treatment within 30 days
* not available for phone follow-up in 3, 7, and 30 days
* requires admission to the hospital
* abnormal mental status.

Ages: 14 Years to 110 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Emergency Medicine Female Patients age ≥14 years of age with a primary urinary complaint.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2022-09-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Resolution of Urinary Tract Infection Symptoms | 3 days (72 hours)
  >80% of patients treated with amikacin will have resolution of urinary tract infection symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Reuben Strayer, MD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-15): https://cdn.clinicaltrials.gov/large-docs/37/NCT05227937/Prot_SAP_000.pdf